CLINICAL TRIAL: NCT04817228
Title: A Prospective Study Performed to Evaluate the Clinical Performance (Debridement), Safety and Pharmacology Effect of EscharEx (EX-02 Formulation) in Patients With Lower Leg Ulcers (VLU and DFU)
Brief Title: A Study to Evaluate the Clinical Performance, Safety and Pharmacology Effect of EscharEx in Patients With Lower Leg Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MediWound Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MW 2020-08-01
Record Dates: First submitted 2021-03-16; First posted 2021-03-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Venous Leg Ulcer; Diabetic Foot Ulcer
MeSH Terms: conditions — Varicose Ulcer; Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EX-02 Gel (Experimental): The powder of EX-02 (8.1 g in each unit) should be reconstituted with 20 g sterile water for injection (WFI) to obtain 5% EX-02. EX-02 5% gel will be topically applied on a wound surface of up to 80 cm2 for 24±3 hours, up to 8 consecutive applications
  Interventions: Drug: EscharEx (EX-02 formulation)

INTERVENTIONS:
Drug: EscharEx (EX-02 formulation) — EscharEx (EX-02 formulation) gel is topically applied on a wound surface of up to 80 cm2 , up to 8 consecutive applications or until a complete debridement is achieved, whichever occurs first.

SUMMARY:
This study will be a multicenter, prospective, open label, one-arm study intended to assess the clinical performance and safety of EX-02 in debridement of lower leg ulcers: Venous Leg Ulcers (VLU) and Diabetic Foot Ulcer (DFU). In addition, the pharmacology effect of EX-02 will be assessed.

Lower leg ulcer size between 2 cm2 and 80 cm2 (surface area).

DETAILED DESCRIPTION:
Up to fifteen (15) adult patients with >50% non-viable tissue (necrotic/ slough/ fibrin) on the ulcer will be enrolled from up to 3 sites.

Each patient will go through the following steps during the trial:

1. Screening and Inform Consent signing - screening visit duration will be up to 1 week and will include: recording demographics, medical history and concomitant medications, vital signs, physical examination, clinical laboratory tests, wound photography and assessments and pain assessment questionnaires. Wound fluid sampling and 3 mm punch biopsy (from the wound edge area) will be taken during screening.
2. Daily visits period (up to 8 daily site visits within up to 14 days), including an additional visit, 48 hrs after last daily visit for wound fluid sampling. During the Daily visits period, the patient will arrive daily to site visits. During each visit, adverse events (AEs), concomitant medications, vital signs, and pain will be assessed and recorded, the wound will be washed, photographed and assessed for wound size and for % of nonviable tissue by clinical assessment. During the daily visits period, the peri-wound will be well protected with topical barrier (e.g zinc oxide paste). For VLU, compression therapy must be used throughout daily visits period.

   The investigator will clinically assess complete debridement, upon achieving a viable wound bed after removal of all non-viable tissue, suitable for initiation of the wound healing stage.

   Patients will be treated with EX-02 for up to 8 applications (up to 8 visits) or until complete debridement is achieved, whichever occurs first. Duration of each application will be 24±3 hours. On weekends occurring during the daily visits period the wound will be dressed with a non-active dressing (e.g. foam).

   Hydrogels as well as methods of active debridement (either surgical, mechanical, biological, enzymatic or other dressings), grafting and V.A.C are not allowed during this period and while daily visits are ongoing.

   Fluid samples will be taken from the EX-02 treated wound before the first treatment and once the wound has reached complete debridement or daily visits completed, whichever occurred first. Punch biopsies from the wound edge will be taken before and at the end of the debridement to assess for biofilm.

   Clinical lab tests and physical examination as well as pain assessments and vital signs will be performed at the end of daily visits period (once the wound has reached complete debridement or daily visits completed, whichever occurred first).

   For patients who achieved complete debridement, wound closure could be considered using grafting/autograft procedure.

   After completion of the daily visits period (either if complete debridement was achieved, or after 8 daily applications were performed) patients will start the weekly follow- up period.
3. Weekly follow- up period (2 visits in 2 weeks) - the 2 weekly follow up period should be performed at the clinical site. During each weekly visit, safety parameters will be recorded (AEs, concomitant medications, pain, vital signs), the wound will be washed, photographed and assessed for wound size and for % of nonviable tissue.

For wounds which did not reach complete debridement during the daily visits period, the investigator should continue to persue complete debridement using surgical or non- surgical debridement tools (SOC), per the investigators discretion.

Compression therapy must be used throughout this period for VLU patients and as determined by investigator to be appropriate for DFU.

The overall duration of the study for each patient will be approximately 4-5 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients, men or women, between 18 and 90 years of age,
2. Patients with a VLU (determined by medical history, physical examination or an ultrasound scan demonstrating venous insufficiency) or DFU (determined by medical history, and physical examination),
3. Wound is present for at least 4 weeks but no longer than 2 years,
4. The necrotic/slough/fibrin non-viable tissue area is at least 50% of wound area (assessed by clinical evaluation),
5. Target wound surface area is in the range of 2-80 cm2,
6. Patient understands the nature of the procedure, is able to adhere to the protocol regimen, and provides a written informed consent prior to any study procedure.

Exclusion Criteria:

1. Patients with more than one leg ulcer, on the leg of the target wound, with an area greater than or equal to 2cm2,
2. Signs of clinically significant infection including purulent discharge, deep-tissue abscess, erysipelas, cellulitis at the surrounding skin, etc.,
3. Severely damaged skin at the per wound (e.g. abrasion, exfoliation) extending >2 cm around the wound's edge,
4. Presence of gangrene, signs of systemic infection, sepsis, or osteomyelitis during screening phase,
5. Clinical suspicion of skin cancer (e.g. BCC, SCC, melanoma, sarcoma), which was not ruled out by biopsy (in this case a biopsy will be performed before screening),
6. Patients suffering from chronic skin disorders (Idiopathic Pruritus, Psoriasis, Panniculitis, Pyoderma Gangrenosum, etc.) that might deteriorate as a result of local trauma or debridement,
7. Wound has sinus tracts or tunnels extending under the skin >2 cm surrounding subcutaneous structures, or penetrating into joint capsule,
8. A significant decrease in the arterial blood flow of the extremity,
9. Patients with pre-enrolment wounds which are covered by eschar heavily saturated with iodine or by silver, silver sulfadiazine (SSD) pseudoeschar (i.e. pseudoeschar as a result of SSD treatment),
10. History of allergy or atopic disease or a known sensitivity to pineapples, papaya, bromelain or papain, as well as known sensitivity to latex proteins (known as latex-fruit syndrome), bee venom or olive tree pollen,
11. Patients with poor nutritional status: albumin < 3.0 g/dl, poorly controlled Diabetes Mellitus (for diabetic patients; HbA1c > 12%), anemia (hemoglobin<8 g/dL), a leukocyte counts < 4,000/ μl or >15000/μl, Neutrophils < 1500/ul, platelets <100,000/μl, abnormal liver function (AST, ALT>2 x upper limit of normal range), total bilirubin > 1.5 mg/dl, renal failure (Cr > 2.5 mg/dl), BMI>45,
12. Patients undergoing renal or peritoneal dialysis,
13. Any condition that would preclude safe participation in the study, e.g. evidence of significant or unstable cardiovascular, pulmonary, liver, hematological, immunological, positive for COVID-19 or neoplastic disease, or any immediate life threatening condition,
14. Recent history (less than 6 months) of myocardial infarction (MI) or concurrent acute injury or disease that might compromise the patient's welfare,
15. Patient is currently receiving, or has received at any time within the past 30 days any medications or treatments known to affect the wound healing processes; these include, chronic systemic steroid intake ( >10 mg/ day) with topical skin changes (i.e. thin, fragile skin with multiple heamatomas or previous laceration history) immuno-suppressive drugs, radiation therapy, immunomodulating medications and chemotherapy,
16. Mentally incapacitated adults who are incapable of giving legal consent (e.g. dementia, psychiatric patients, etc.),
17. Concurrent use of non-approved drugs or alcohol abuse,
18. Pregnant women (positive pregnancy test) or nursing mothers,
19. Exposure to investigational intervention within 3 months prior to enrollment, or anticipated participation in another investigational drug trial or other intervention trial, while enrolled into the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Incidence of complete debridement | up to 14 days
  Incidence of complete debridement assessed clinically
Time to complete debridement | up to 14 days
  Time to complete debridement assessed clinically
Change from baseline in wound fluid biomarkers | up to 14 days
  Wound healing biomarkers (MMP2, MMP9, HNE, PDGF, IL8, TNFR1) distribution in wound fluid will be compared before and after completion of treatment
Change from baseline in wound biofilm presence before and after treatment | up to 14 days
  Biofilm presence in wound will be compared before and after completion of treatment, using punch biopsy from wound

CONTACTS AND LOCATIONS:
Overall Officials: Lior Rosenberg, Prof., Study Chair — MediWound Ltd
Locations (3):
- United States (3):
  - Barry University foot and ankle institute, Tamarac, Florida
  - Clinical Research Medical Center, LLC, Las Vegas, Nevada
  - University of North Carolina, Chapel Hill, North Carolina